CLINICAL TRIAL: NCT07239453
Title: An Open-Label, Randomized, Single Oral Dose, Two-Sequence, Two-Period, CrossovSer Bioequivalence Study of "DA-2902" and "DA-2902-R" in Healthy Adults Under Fed Conditions
Brief Title: Clinical Trial of Comparing DA-2902 and DA-2902-R in Healthy Adult Subjects
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA2902_BE_I
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Infective Disorder
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental)
  Interventions: Drug: DA-2902; Drug: DA-2902-R
- Sequence B (Experimental)
  Interventions: Drug: DA-2902; Drug: DA-2902-R

INTERVENTIONS:
Drug: DA-2902 — single dose administration (DA-2902 one tablet once a day)
Drug: DA-2902-R — single dose administration (DA-2902-R one tablet once a day)

SUMMARY:
This study is to compare pharmacokinetics and safety profiles of DA-2902 and DA-2902-R in healthy adult subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* BMI between 18 and 30 kg/m2
* Body weight: Male≥50kg, Female≥45kg
* Subjects who have signed an informed consent themselves after receiving detailed explanation about clinical study

Exclusion Criteria:

* Subjects with clinically significant medical history
* Subjects with history of drug abuse or addicted
* Subjects with allergy or drug hypersensitivity

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
AUCt | pre-dose ~ 72 hr of pose-dose
Cmax | pre-dose ~ 72 hr of post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- CHA University Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea